CLINICAL TRIAL: NCT00884585
Title: Efficacy and Safety Study of Cyclosporine 0.010% to Treat Atopic Keratoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192371-016
Record Dates: First submitted 2009-04-17; First posted 2009-04-21 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Atopic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine Ophthalmic Solution (COS) followed by COS (Experimental): Cyclosporine ophthalmic solution 0.010% administered 4 times a day to the qualified eye(s) for up to 12 months; at Month 9 the dose may be adjusted to 2 times a day.
  Interventions: Drug: Cyclosporine 0.010%
- Placebo followed by COS (Other): Placebo (cyclosporine vehicle) administered 4 times a day to the qualified eye(s) for 3 months followed by cyclosporine ophthalmic solution 0.010% up to 9 additional months; at Month 9 the dose may be adjusted to 2 times a day.
  Interventions: Drug: Cyclosporine Vehicle; Drug: Cyclosporine 0.010%

INTERVENTIONS:
Drug: Cyclosporine Vehicle — Placebo (cyclosporine vehicle) administered 4 times a day to the qualified eye(s) for 3 months.
  Arms: Placebo followed by COS
Drug: Cyclosporine 0.010% — Cyclosporine ophthalmic solution 0.010% administered 4 times a day to the qualified eye(s) for up to 12 months; at Month 9 the dose may be adjusted to 2 times a day.

SUMMARY:
This study evaluates the efficacy and safety of Cyclosporine 0.010% eye drops in the treatment of Atopic Keratoconjunctivitis (chronic and severe inflammation of the eye). The study consists of a double-masked phase, and open-labeled phase, and an open-labeled maintenance phase. For the first 3 months of the study, patients will receive either masked Cyclosporine 0.010% eye drops or vehicle four times daily; for the next 6 months, patients may receive open-labeled Cyclosporine 0.010% eye drops four times daily. At month 9, patients who are in remission, will be re-randomized to receive either open-labeled Cyclosporine 0.010% eye drops four times daily or twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of Atopic Keratoconjunctivitis (chronic and severe inflammation of the eye)
* Be on stable doses of your current AKC medications for at least 2 weeks

Exclusion Criteria:

* You have used contact lenses within 48 hours of Day 1 or think you may have to wear contact lenses during the study
* You are pregnant, breastfeeding, or planning to become pregnant during the study
* You have used a calcineurin inhibitors (e.g. topical tacrolimus or topical pimecrolimus) on or around your eyes including eyelids within 4 weeks

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (12):
- Bakersfield, California, United States
- Randwick, New South Wales, Australia
- Ottawa, Ontario, Canada
- Prague, Czechia
- Dijon, Burgundy, France
- Munich, Bavaria, Germany
- Bangalore, Karnataka, India
- Tel Aviv, Israel
- Rome, Italy
- Wellington, New Zealand
- Valladolid, Spain
- Newcastle upon Tyne, Tyne and Wear, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol defined pre-specified criteria, both eyes could qualify for treatment. However, only one eye was designated as the study eye.
Period: Double-Masked Phase (Day 1-Month 3)
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo Followed by COS
Started | 89 | 87
Completed | 79 | 83 (All placebo patients who completed the double-masked phase received COS in the open-label phase.)
Not Completed | 10 | 4
Period: Open-Label Phase (Months 3-9)
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo Followed by COS
Started | 162 (All patients who completed the double-masked phase received COS in the open-label phase.) | 0 (All placebo patients who completed the double-masked phase received COS in the open-label phase.)
Completed | 147 | 0
Not Completed | 15 | 0
Period: Open-Label Maintenance (Months 9-12)
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo Followed by COS
Started | 147 | 0
Completed | 144 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo Followed by COS | Total
Number analyzed (Participants) | 89 | 87 | 176
Age, Customized [Number; unit: Participants]
  <18 years | 7 | 8 | 15
  18 to <30 years | 15 | 13 | 28
  30 to <50 years | 32 | 38 | 70
  50 to <65 years | 27 | 22 | 49
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 39 | 85
  Male | 43 | 48 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders
Description: Treatment responders are defined as patients with a ≥ 1 grade improvement from baseline in punctate corneal staining score and a ≥ 4 grade improvement from baseline in composite symptom score in the study eye. The punctate corneal staining score is assessed on a scale of 0 to 5 (0 is ≤2 dots and 5 is >316 dots (approximately) or ulcer/erosion). The composite symptom score is based on 5 symptoms (itching, tearing, ocular discomfort, photophobia, mucous discharge). The composite symptom score (0 to 15) is the sum of 5 symptoms (each symptom is assessed on a scale of 0=absent to 3=severe).
Time Frame: Baseline, Month 2
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Groups:
- Placebo: Placebo (cyclosporine vehicle) administered 4 times a day to the qualified eye(s) for 3 months.
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo
Number analyzed (Participants) | 89 | 87
Percentage of Patients | 21.3 | 17.2

2. Secondary Outcome: Percentage of Punctate Corneal Staining Responders
Description: Punctate corneal staining responders defined as patients achieving a punctate corneal staining score of 0 or 1 in the study eye. Punctate corneal staining is assessed on a scale of 0 to 5 where 0 is ≤2 dots, 1 is >2 dots but ≤ 10 dots, 2 is > 10 dots but ≤ 32 dots, 3 is > 32 dots but ≤ 100 dots (approximately), 4 is > 100 dots (approximately) but ≤ 316 dots (approximately), and 5 is >316 dots (approximately) or ulcer/erosion.
Time Frame: Month 2
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo
Number analyzed (Participants) | 89 | 87
Percentage of Patients | 24.7 | 23.0

3. Secondary Outcome: Percentage of Patients With an Improvement in the Composite Symptom Score
Description: Composite symptom score improvement is defined as a 4 or more grade decrease from baseline in composite symptom score in the study eye. The composite symptom score is based on 5 symptoms (itching, tearing, ocular discomfort, photophobia, mucous discharge). Each of the 5 symptoms is assessed on a scale of 0=absent to 3=severe. The composite symptom score is the sum of all 5 individual symptom scores, where 0 is no symptoms and 15 is the most severe symptoms.
Time Frame: Baseline, Month 2
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo
Number analyzed (Participants) | 89 | 87
Percentage of Patients | 30.3 | 28.7

4. Secondary Outcome: Percentage of Patients With an Improvement in the Punctate Corneal Staining Score
Description: Punctate corneal staining improvement is defined as a 1 or more grade decrease from baseline in the study eye. The punctate corneal staining score is assessed on a scale of 0 to 5 where 0 is ≤2 dots, 1 is >2 dots but ≤ 10 dots, 2 is > 10 dots but ≤ 32 dots, 3 is > 32 dots but ≤ 100 dots (approximately), 4 is > 100 dots (approximately) but ≤ 316 dots (approximately), and 5 is >316 dots (approximately) or ulcer/erosion.
Time Frame: Baseline, Month 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo
Number analyzed (Participants) | 89 | 87
Percentage of Patients | 42.7 | 42.5

ADVERSE EVENTS:
Description: The Safety Population was used for all adverse event (AE)/serious adverse event (SAE) reporting. All patients in the safety population received at least 1 dose of study medication.
Arm/Group | Cyclosporine Ophthalmic Solution (COS) Followed by COS | Placebo
Serious Adverse Events (participants affected / at risk) | 11/171 | 3/87
Other Adverse Events (participants affected / at risk) | 44/171 | 16/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine Ophthalmic Solution (COS) Followed by COS (N=171) | Placebo (N=87)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infectious Mononucleosis (Infections and infestations) | 1 | 0
Prostatic Specific Antigen Increased (Investigations) | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine Ophthalmic Solution (COS) Followed by COS (N=171) | Placebo (N=87)
Allergic Keratitis (Eye disorders) | 24 | 10
Blepharitis (Eye disorders) | 10 | 3
Punctate Keratitis (Eye disorders) | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.